CLINICAL TRIAL: NCT05506228
Title: How Are the Muscles Affected in Cerebral Palsy? A Study of Muscle Biopsies Taken During Orthopaedic Surgery of Children With Cerebral Palsy and Typically Developed Children (Control).
Brief Title: How Are the Muscles Affected in Cerebral Palsy? A Study of Muscle Biopsies Taken During Orthopaedic Surgery.
Acronym: CPTDBiopsy
Status: Recruiting | Type: Observational
Sponsor: Eva Ponten (Other Government)
Responsible Party: Sponsor-Investigator, Eva Ponten, Principal Investigator, Region Stockholm
Organization: Region Stockholm (Other Government)
Other Study IDs: CP muskel OP + kontr
Record Dates: First submitted 2022-07-27; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Palsy; Muscle; Muscle Contracture; Muscle Spasticity
Keywords: Cerebral Palsy; Upper Limb; Lower Limb; Muscle Biopsy; Plasma
MeSH Terms: conditions — Cerebral Palsy; Contracture; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Muscle and tendon biopsies. Blood samples for serum and plasma analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebral Palsy (CP) / Acquired Brain Injury (ABI): Children and adolescents with cerebral palsy and acquired brain injury.
  Interventions: Other: No intervention
- TD (Typically Developed): Typically developed children and adolescents.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
* Cerebral palsy (CP) is a motor disorder caused by an injury to the immature brain. Even though the brain damage does not change, children with CP will have progressively weaker, shorter and stiffer muscles that will lead to contractures, bony deformations, difficulty to walk and impaired manual ability. An acquired brain injury (ABI) later during childhood, such as after a stroke or an injury, will result in similar muscle changes, and will therefore also be included in this study. For simplicity, these participants will in this text be referred to as having CP.
* The mechanism for the muscle changes is still unknown. Contractures and the risk for the hips to even dislocate is now treated by tendon lengthening, muscle release and bony surgery. During these surgeries muscle biopsies, tendon biopsies and blood samples will be taken and compared with samples from typically developed (TD) children being operated for fractures, knee injuries, and deformities. The specimens will be explored regarding inflammatory markers, signaling for muscle growth, signaling for connective tissue growth and muscle and tendon pathology. In blood samples, plasma and serum, e.g. pro-inflammatory cytokines and the cytoprotective polypeptide humanin will measured, and will be correlated to the amount humanin found in muscle. With this compound information the mechanism of contracture formation may be found, and hopefully give ideas for treatment that will protect muscle and joint health, including prevention of hip dislocation and general health.
* The results will be correlated to the degree of contracture of the joint and the severity of the CP (GMFCS I-V, MACS I-V).
* By comparing muscle biopsies from the upper limb with muscle biopsies from the lower limb, muscles that are used in more or less automated gait will be compared to muscles in the upper limb that are used more voluntarily and irregularly.
* Muscles that flex a joint, often contracted, will be compared with extensor muscles from the same patient. Fascia, aponeurosis and tendon will also be sampled when easily attainable.

DETAILED DESCRIPTION:
* Cerebral palsy (CP) is a motor disorder caused by an injury to the immature brain. Even though the brain damage does not change, children with CP will have progressively weaker, shorter and stiffer muscles that will lead to contractures, bony deformations, difficulty to walk and impaired manual ability. An acquired brain injury (ABI) later during childhood, such as after a stroke or an injury, will result in similar muscle changes, and will therefore also be included in this study. For simplicity, these participants will in this text be referred to as having CP.
* The mechanism for the muscle changes is still unknown. Contractures and the risk for the hips to even dislocate is now treated by tendon lengthening, muscle release and bony surgery. During these surgeries muscle biopsies, tendon biopsies and blood samples will be taken and compared with samples from typically developed (TD) children being operated for fractures, knee injuries, and deformities. The specimens will be explored regarding inflammatory markers, signaling for muscle growth, signaling for connective tissue growth and muscle and tendon pathology. In blood samples, plasma and serum, e.g. pro-inflammatory cytokines and the cytoprotective polypeptide humanin will be measured and correlated to the amount humanin found in muscle. With this compound information the mechanism of contracture formation will hopefully be found and give ideas for treatment that will protect muscle and joint health including prevention of hip dislocation and general health.
* Research questions:

Contracture formation in CP is caused by:

Stiffer muscle/tendon complex? Is there more extracellular matrix around the muscle fiber bundles in CP? Are there pathological intramuscular aponeuroses and tendons? Reduced muscle growth? Are the satellite cells fewer and less active in CP? Is the ribosome number and function affected? Are pro-inflammatory cytokines increased, diminishing growth?

Muscle weakness in CP is caused by impaired metabolic function, caused by:

Fewer mitochondriae? Less mitochondrial ribosomes? Higher percentage of the faster and fatigable myosin MHCIIX? More developmental myosins (neonatal and embryonic myosin)? Decreased PGC-1α?

• Blood samples: Will there be increased expression of pro-inflammatory cytokines, correlating to cytokine expression in muscle and to muscle pathology? Is humanin levels in plasma correlated to muscle levels?

* Muscle samples and tendon samples will be taken during clinically indicated and planned orthopaedic surgery from muscles that are easily exposed from the incisions needed for the primary surgery. Muscle samples 3x3x8 mm from 2-8 different muscles will be taken in such a way that there will be no diminished clinical function. Tendon samples 3x3x3 mm will be taken so that no biomechanical damage occurs. The samples are snap frozen and are stored in -80°C for later analyses. Biopsies are also put fresh in Allprotect (Qiagen) which stabilizes DNA, RNA and proteins, and are kept in a refrigerator for later analyses with e.g. ELISA and PCR.
* The results will be correlated to the degree of contracture of the joint and the severity of the CP (GMFCS I-V, MACS I-V).
* By comparing muscle biopsies from the upper limb with muscle biopsies from the lower limb, muscles that are used in more or less automated gait can be compared to muscles in the upper limb that are used more voluntarily and irregularly.
* Muscles that flex a joint, often contracted, will be compared with extensor muscles from the same patient. Fascia, aponeurosis and tendon will also be sampled when easily attainable.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents undergoing clinically needed orthopaedic surgery
* with Cerebral Palsy or Acquired Brain Injury
* Typically developed children and adolescents (control)

Exclusion Criteria:

* for CP/ABI: Progressive neurological disease, other metabolic or muscle disease
* for TD (Control): Cerebral Palsy, Acquired Brain injury, other metabolic or muscle diseases

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients who are scheduled for clinically needed orthopaedic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2002-01-15 (Actual); Primary Completion 2032-12-15 (Estimated); Study Completion 2033-12-15 (Estimated)

PRIMARY OUTCOMES:
Muscle/tendon morphology | 2002- 2027
  morphology classification
Muscle metabolism | 2002- 2027
  NADH staining classification
Fiber area | 2002- 2027
  um 2, square micrometer

SECONDARY OUTCOMES:
Clinical data, Contracture | Pre-OP
  degrees

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Pontén, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided